CLINICAL TRIAL: NCT01741103
Title: Effect of Sitagliptin on Glycemic Control, Post-prandial Glucagon, and Inflammation in Type 1 Diabetics
Brief Title: Sitagliptin in Type I Diabetic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding was for 1 year to a fellow who graduated in early stages of enrollment. While 6 patients were enrolled, many patients didn't finish the study and therefore little data was collected and no results will be entered.
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, Clinical Professor of Medicine, Kaleida Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1957
Record Dates: First submitted 2011-09-27; First posted 2012-12-04 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental)
  Interventions: Drug: sitagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sitagliptin — sitagliptin 100mg by mouth once a day for 12 weeks
  Other Names: Januvia/Sitagliptin 100mg
  Arms: Sitagliptin
Drug: Placebo — Take one by mouth daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of sitagliptin on overall blood glucose concentrations in Type I Diabetic subjects. The study also aims to evaluate post meal glucagon concentrations in Type I Diabetic subjects (a possible mechanism of reduced blood glucose concentrations) and indices of oxidation stress in the plasma of these subjects.

DETAILED DESCRIPTION:
The hypothesis is that Sitagliptin will improve overall blood glucose, fasting blood glucose, and glycemic excursions in patients with Type I Diabetes. In addition, sitagliptin will likely suppress indices of oxidative stress in patients. The study will investigate proposed mechanisms of improved glucose concentrations, including enhanced effect of endogenous GLP-1 and suppression of glucagon.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult, aged 18 to 70 years
2. Type 1 Diabetes Mellitus for 6 months or more, as established by medical history
3. Current treatment with multiple injections of insulin (at least 4) or CSII (continuous subcutaneous insulin infusion or insulin pump) therapy for at least 3 months prior to screening visit; and using the same insulin during the last 1 month
4. HbA1c ≤ 8.5%
5. Subjects should routinely practice at least 2-4 blood glucose measurements per day
6. BMI ≤ 35 kg/m2
7. Subject must be able and willing to perform self-blood glucose monitoring and accept wearing a continuous glucose monitor for 3 days at the start and 3 days at the end of the study
8. Subjects must be willing to complete study visits per study protocol
9. Able to speak, read, and write English

Exclusion Criteria:

1. Type 1 Diabetes Mellitus for less than 6 months
2. Coronary Event or procedure (myocardial infarction, unstable angina, coronary artery bypass surgery, or coronary angioplasty) in the previous 4 weeks
3. Any other life-threatening, non-cardiac disease
4. Pregnant or intends to become pregnant during the course of the study
5. Severe unexplained hypoglycemia that required emergency treatment over the past 3 months
6. History of hemoglobinopathies
7. Post-renal transplantation, currently undergoing dialysis, creatinine of >1.5mg/dl or a calculated creatinine clearance of <50 mL/min.
8. Have extensive skin changes/diseases that inhibit wearing the sensor on normal skin
9. Subjects who have an allergy to medication being used
10. Current participation in another study protocol
11. History of autonomic neuropathy or gastroparesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
change from baseline in mean glucose concentrations | baseline and 3 months
  The primary endpoint of the study is to detect the change from baseline in mean glucose concentrations as measured by both HbA1c, and mean glucose over the three days of continuous glucose monitoring.

SECONDARY OUTCOMES:
Glycemic changes | baseline and 3 months
  Glycemic changes including standard deviations of the glycemic levels, fructosamine, and the duration of time spent in hyperglycemia and hypoglycemia.
Post meal hyperglycemia | baseline and 3 months
  Post meal hyperglycemia will be measured as area under the curve (AUC).
Changes in post prandial glucose, glucagon, insulin, c-peptide, DPP-IV, GIP and, GLP-1 concentrations following meal challenge. | baseline and 3 months
Changes in NF kappa B in the fasting state. | baseline and 3 months
Change in NFkappaB following meal challenge. | baseline and 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — Kaleida Health and University at Buffalo
Locations (1):
- 115 Flint Road, Williamsville, New York, United States